CLINICAL TRIAL: NCT01126632
Title: Will Cap-Assisted Colonoscopy Improve Performance of Colonoscopy: A Randomized Clinical Trial
Acronym: CAC
Status: Withdrawn | Type: Observational
Why Stopped: Caps became unavailable by manufacturer
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: CAC Study
Record Dates: First submitted 2010-05-15; First posted 2010-05-20 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Colonoscopy
Keywords: Colonoscopy

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cap Assisted Colonoscopy: Patients receiving colonoscopies where scope is fitted with cap
- Standard Colonoscopy: Patients receiving standard colonoscopy without the cap on the scope

SUMMARY:
Observing the effects of an Olympus cap on the visibility and in adenoma detection during colonoscopy.

DETAILED DESCRIPTION:
To see if Colonoscopy with the CAP is able to give more visibility and to see if detection rate for adenomas, polyps are easier to detect.

ELIGIBILITY:
Inclusion Criteria:

* Patients already booked for a colonoscopy

Exclusion Criteria:

* History of Colorectal Cancer
* Severe colitis
* Cancer
* poor bowel prep

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Endoscopy Clinic- Patients already receiving colonoscopies
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
cap-assisted colonoscopy compared visibility with standard colonoscopy | 4 months
  Propose to perform a randomized controlled trial comparing cap-assisted colonoscopy with the standard colonoscopy to assess visibility. To see if it is easier to detect polyps, adenomas with the cap than without. This is standard procedure. Just comparing if it is better to use the cap during colonoscopy.

SECONDARY OUTCOMES:
Polyp detection rate | 4 months
  Number of Polyps detected per procedure using the cap. To see if it is more visible.
Adenoma Detection | 4 months
  number of adenomatous polyps detected per procedure. To see if it is more visible using the cap as to not using the cap.
Advanced lesion detection rate | 4 months
  (number of advanced lesions per procedure) defined as lesions with high-grade dysplasia, greater than 1 cm. size. To see if it is more visible using the cap as to not using the cap.
Cecal Intubation Rate | 4 months
  Time to cecum
Total time for colonoscopy | 4 months
Complication Rate | 4 months
  Amount of complications during colonoscopies
Procedure indication | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Donald G MacIntosh, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Study was terminated

REFERENCES:
- [Result] Lee YT, Lai LH, Hui AJ, Wong VW, Ching JY, Wong GL, Wu JC, Chan HL, Leung WK, Lau JY, Sung JJ, Chan FK. Efficacy of cap-assisted colonoscopy in comparison with regular colonoscopy: a randomized controlled trial. Am J Gastroenterol. 2009 Jan;104(1):41-6. doi: 10.1038/ajg.2008.56. PMID 19098847